CLINICAL TRIAL: NCT01946867
Title: A Phase I Dose-Escalation/Dose Expansion Study Of NBTXR3 Activated By Intensity Modulated Radiation Therapy In Patients With Locally Advanced Squamous Cell Carcinoma Of The Oral Cavity Or Oropharynx
Brief Title: NBTXR3 and Radiation Therapy in Treating Patients With Locally Advanced SCC of the Oral Cavity or Oropharynx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanobiotix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBTXR3-102; ID RCB: 2013-A00706-39 (Other: Other)
Record Dates: First submitted 2013-09-10; First posted 2013-09-20 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Head and Neck Cancer
Keywords: Oral cavity Cancer; Oropharynx Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms; Oropharyngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: This study consists of two parts: Dose Escalation and Dose Expansion. This phase I is an open-label non-randomized, dose-escalation/dose expansion study of safety and tolerability evaluation of NBTXR3, administered as an intratumoral implantation by injection, activated by intensity modulated radiation therapy (IMRT), in patients with locally advanced squamous cell carcinoma of the oral cavity or oropharynx.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NBTXR3 IntraTumoral injection (IT) (Experimental): Single intratumor injection
  Interventions: Device: NBTXR3 activated by IMRT

INTERVENTIONS:
Device: NBTXR3 activated by IMRT

SUMMARY:
RATIONALE: Cancers of the oral cavity represent 30% of head and neck carcinomas in the western world. The oropharynx is the posterior continuation of the oral cavity and connects with the nasopharynx (above) and laryngopharynx (below). It is also a frequent site of primary head and neck cancers. These structures play a crucial role in swallowing, breath and speech. Locally advanced oropharyngeal cancers can obstruct the air flow or infiltrate muscles or nerves, which significantly disturb local functions. The incidence of Head and Neck Squamous Cell Cancer in patients older 65 years is high, 47% occurred in this population as recorded by the Surveillance, Epidemiology, and End Results registries in the United States. Regarding the therapeutic strategies, the association of radiotherapy with chemotherapy or biologics has demonstrated significant improvement of outcomes with the drawback of higher toxicity, or as demonstrated by 2 meta-analyses, without survival improvement in older patients. NBTXR3 and radiation therapy may increase the cancer cell killing and complete tumor shrinkage allowing a definitive treatment and preservation of local structures and functions in patients older 65 years, who cannot receive cisplatin.

DETAILED DESCRIPTION:
Patients will receive a single administration of NBTXR3 on day 1,as an intratumor injection, followed by Intensity Modulated Radiation Therapy starting 24 hours later (Day 2), and up to completion of 7 weeks, i.e. 70 Grays, 2Grays/fraction. Patients whose tumor has completely shrunk will be followed for the post-radiotherapy evaluation up to the End of Treatment visit. Those patients whose tumor has not shrunk more than 50% of the baseline size, will stop the radiotherapy and may have a salvage tumor surgery. Then, all patients will be followed every 8 weeks, for the safety evaluation and cancer disease status until the end of the study.

ELIGIBILITY:
Inclusion criteria:

* Patients aged ≥ 70 years old, or
* Patients aged ≥ 65 years old and < 70 years old who are unable to receive cisplatin, or
* Patients who have contraindication to cisplatin or that are intolerant to cisplatin or cetuximab or that cannot receive the combination of chemoradiation, regardless the age
* Histologically or cytologically confirmed squamous cell carcinoma (SCC) of the oral cavity or oropharynx
* T3 or T4 primary tumor or Stage III or IVA according to AJCC guidelines (8th Edition, 2018)
* No evidence of distant metastatic disease, as determined by a negative PET scan or CT scan
* Clinically eligible for intratumor implantation by injection
* Karnofsky Performance Status ≥ 70
* Adequate function of Bone marrow:

  * White Blood Cell (WBC) > 3.0 x 10^9/L
  * Absolute neutrophil count (ANC) > or = 1.0 x 10^9/L
  * Platelet count > or = 100 x 10^9/L
  * Hemoglobin > or = 9.0 g/dL
* Adequate function of Kidney:

  o Creatinine < or = 3.0 x ULN or creatinine clearance > or = 30 mL/min/1.73m²
* Adequate function of the liver:

  * AST < or = 5 x ULN
  * ALT < or = 5 x ULN
  * Bilirubin < or = 1.5 x ULN
* Negative pregnancy test ≤ 7 days of NBTXR3 injection in all females of child-bearing potential

Exclusion Criteria:

* Written Informed Consent not obtained, signed and dated
* Prior radiotherapy to any area within the planned radiotherapy field
* Tumor-related dyspnea
* Tumor ulceration which implies vascular risk
* Non measurable disease as defined by RECIST criteria
* History of stroke, CABG, or significant blockage of carotid arteries or coronary arteries or current blockage of coronary or carotid arteries equal to or in excess of 50% blockage
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active severe infection, symptomatic congestive heart failure, acute coronary syndrome, etc.
* Medical history of life-threatening ventricular arrhythmia
* Prior or concurrent non-head and neck malignancies, excluding adequately treated basal or squamous cell cancer of the skin, and in situ cervical cancer, and any other cancer from which the subject has been cancer free for 5 years
* Concurrent treatment with any other anticancer therapy, including chemotherapy, immunotherapy, targeted therapy, gene therapy, or patients planning to receive these treatments during the study
* Patients unable to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures or those with severe psychiatric illness/social situations that would limit compliance with study requirements
* Patients participating in another clinical investigation at the time of signature of the informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-01-03 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Incidence of DLTs and determination of the Recommended Phase 2 Dose | 12 months
  The incidence of early DLTs (early adverse effects related to NBTXR3, as an intratumor injection, activated by IMRT)
Dose Escalation: Determination of the Recommended Phase 2 Dose | 12 months
  The recommended Phase II dose (RD) of NBTXR3 administered as intratumor injection, activated by Intensity Modulated Radiation Therapy (IMRT)
Dose Expansion: Overall Response Rate | 12-24 months
  The Objective Response Rate (ORR) of the primary tumor, by imaging according to RECIST 1.1
Dose Expansion: Complete Response Rate | 12-24 months
  The Complete Response Rate (CRR) of the primary tumor, by imaging according to RECIST 1.1

SECONDARY OUTCOMES:
Dose Escalation: Objective Response Rate (ORR) of the primary tumor | 12-24 months
  The Objective Response Rate (ORR) of the primary tumor, by imaging according to RECIST 1.1
Dose Escalation: Complete Response Rate | 12 months
  The Complete Response Rate (CRR) of the primary tumor, by imaging according to RECIST 1.1
Dose Expansion: Local Progression Free Survival | 12-24 months
  Local Progression Free Survival (LPFS) defined as any recurrence at the site of the primary tumor
Dose Expansion: Progression Free Survival | 12-24 months
  Progression Free Survival (PFS) defined as the time to any progression at the site of the primary tumor, in regional lymph nodes and/or distant metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Christophe LE TOURNEAU, MD-PhD, Principal Investigator — Institut Curie Paris France
Locations (20):
- France (8):
  - Centre Francois Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Hôpital La Timone, Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - CHU Pontchaillou, Rennes
  - Institut de Cancérologie de la Loire Lucien Neuwirth, Saint-Priest-en-Jarez
  - Institut Gustave Roussy, Villejuif
- Hungary (2):
  - Hungarian Defense Forces Hospital, Budapest
  - National Institute of Oncology, Budapest
- Poland (5):
  - Centrum Onkologii - Instytut im. M. Skłodowskiej- Curie, Oddział w Gliwicach, Gliwice
  - Świętokrzyskie Centrum Onkologii Samodzielny Publiczny Zakład Opieki Zdrowotnej W Kielcach, Kielce
  - Centrum Onkologii Ziemi Lubelskiej im. Św. Jana z Dukli, Lublin
  - NU-MED, Provita Prolife, Tomaszów Mazowiecki
  - Nu-Med Centrum Diagnostyki I Terapii Onkologicznej Zamość Spółka Z Ograniczoną Odpowiedzialnością, Zamość
- Spain (5):
  - Institut Catala d'Oncologia Hospital, Barcelona
  - Vall d'Hebron Hospital, Barcelona
  - Hospital Fundación Jimenez Diaz, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Hospital Universitario Regional de Malaga, Málaga

REFERENCES:
- [Derived] Le Tourneau C, Liem X, Nguyen F, Deraedt S, Salas S, Calugaru V, Serrahima MP, Wong Hee Kam S, Hoffmann C, Lesnik M, Blanchard P, Poissonnet G, Bozec A, Saada-Bouzid E, Jegoux F, Castelli J, Devisetty K, Lelonge Y, Jadaud E, Houdas L, Debard A, Vivar OI, Finzi L, Serra A, Linares I, Arranz Obispo C, Thariat J, Rambeau A, Fakhry N, Santini L, Giralt J, Brana Garcia I, Barba MS, Gorphe P, Helfferich F, Herczeg A, Papai Z, Fijuth J, Takacsi-Nagy Z. Intratumoral Radioenhancer Nanoparticle NBTXR3 Followed by Radiotherapy in Head and Neck Cancer: A Phase 1 Dose-Expansion Nonrandomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2026 Jan 29:e254939. doi: 10.1001/jamaoto.2025.4939. Online ahead of print. PMID 41609775
- [Derived] Hoffmann C, Calugaru V, Borcoman E, Moreno V, Calvo E, Liem X, Salas S, Doger B, Jouffroy T, Mirabel X, Rodriguez J, Chilles A, Bernois K, Dimitriu M, Fakhry N, Hee Kam SW, Le Tourneau C. Phase I dose-escalation study of NBTXR3 activated by intensity-modulated radiation therapy in elderly patients with locally advanced squamous cell carcinoma of the oral cavity or oropharynx. Eur J Cancer. 2021 Mar;146:135-144. doi: 10.1016/j.ejca.2021.01.007. Epub 2021 Feb 16. PMID 33607477